CLINICAL TRIAL: NCT02936050
Title: The Use of Ultrasound Diagnostics for Clinical Decision Making at Remote Locations - Data From an Outpatient Heart Failure Clinic
Brief Title: Telemedicine for Ultrasound Support in Nurse-based Outpatient Heart Failure Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Nord-Trøndelag HF (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LH_2016-1
Record Dates: First submitted 2016-09-26; First posted 2016-10-18 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Heart Failure
Keywords: Echocardiography; Telemedicine; Nurses; Decision support; eHealth
MeSH Terms: conditions — Heart Failure | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Other): Experimental: Addition of diagnostic ultrasound performed by nurses at the outpatient heart failure clinic. Interpretation by specialist per telemedicine.
  No Control arm
  Interventions: Procedure: Diagnostic ultrasound

INTERVENTIONS:
Procedure: Diagnostic ultrasound — All participants will be examined by diagnostic ultrasound by nurses for the assessment of the Cardiac size and function, and for volumic state. Transmission of the ultrasound recordings by telemedicine and interpretation by specialist in echocardiography and heart failure. All participants will then be examined by reference imaging in specific ultrasound laboratories.
  Other Names: Echocardiography

SUMMARY:
The cost related to management of heart failure is significant, both with respect to the financial costs and the suffer of patients. Still as much as 50% of heart failure patients are readmitted within 6 months after hospitalization for decompensated heart failure.

Specialized nurses have a growing role in diagnostics and follow-up of outpatient HF patients, and adding ultrasound diagnostics to the nurses consultations may improve care. In heart failure patients the use of ultrasound as a tool for assessing volume status and guidance of diuretic therapy are promising. Aim of the study is to evaluate the feasibility and reliability of echocardiographic acquisitions by heart failure nurses to assess cardiac function indices and assess volume status in outpatient heart failure clinics combined with a telemedicine approach for near real-time interpretation of the recordings by a cardiologist specialized in echocardiography and heart failure at a remote location.

DETAILED DESCRIPTION:
The worsening heart failure epidemic is a significant driver of health care expenditure with increasing costs, lost productivity and increased suffer of patients. Thus, there important to develop strategies to improve heart failure care and reduce hospital readmissions. Some progress in heart failure management has been made with new drug therapies and remote monitoring of patients with heart failure.

This project aims to provide data which may add to the existing literature regarding the use of telemedicine for safe transfer of ultrasound data of relatively inexperienced users for qualitative and quantitative interpretation by experts at a different location. The authors will study whether diffusion of focused cardiac ultrasound to outpatient heart failure clinics with support of cardiologist provided by telemedicine is feasible and provides reliable data. Firstly, the investigators will study the use of high-end ultrasound machines connected to a wired broadband network with a CE-classified software providing safety and anonymization of all transferred data.

This project could be of significant importance for further support for widening the use of ultrasound diagnostics, even when the expert is not at the same location as the health-care provider performing the ultrasound acquisition. For the patients this may allow for better and faster diagnostics, and thus treatment. For the health-care system this may both improve quality of diagnostics and therapy, and be cost-saving as well. Lastly, this could make the way for further innovations which again can improve diagnostics and thus therapy.

Aims

1. To study the feasibility of implementing focused echocardiography and ultrasound examinations to assess volume status in a heart failure clinic where the caregiving nurses acquire the ultrasound images but have access to the near real-time interpretation by the cardiologist only by telemedicine.
2. To study the reliability of the measurements of cardiac size and function indices in ultrasound recordings acquired by heart failure nurses, provided to another location for interpretation by cardiologists by telemedicine, in comparison to reference imaging.
3. To study the clinical influence of implementing ultrasound examinations performed by nurses to assess volume status and cardiac function at outpatient heart failure clinics when the support and collaboration with the specialist is available by telemedicine only.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure patients at the outpatient heart failure clinic at Levanger Hospital, which have consented to participate in the study.

Exclusion Criteria:

* As for inclusion, when the patient is not able to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Reliability of diagnostic ultrasound examinations using support by telemedicine | Reliability will be tested on day 0 (time of study inclusion)
  Reliability (accuracy) will be tested with C-statistics of ultrasound performed by nurses at an outpatient heart failure clinic, with interpretation by telemedicine support of cardiologist compared to Reference imaging by specialists in cardiology

SECONDARY OUTCOMES:
Feasibility of echocardiography performed by nurses with support by telemedicine | Feasibility will be tested on day 0 (time of study inclusion)
  Feasibility, as the proportion of recordings, of echocardiographic images with telemedicine interpretation of the echocardiographic recordings. Specified will we evaluate the proportion of exams that is successfully recorded by the nurses, then transmitted by and, at last, interpretated by telemedicine approach.
Time use of echocardiography performed by nurses with support by telemedicine | Feasibility will be tested on day 0 (time of study inclusion)
  Time used for the sum of recording of echocardiographic images by the nurses, uploading for transferral and, at last, interpretation by telemedicine approach.
Quality of echocardiography performed by nurses with support by telemedicine | Quality will be tested on day 0 (time of study inclusion)
  Evaluation of the quality of recordings of echocardiographic images obtained by the nurses as a semiquantitative score reflecting the whole examination compared to the reference images by the cardiologist.
Classification of type of heart failure by echocardiography by nurses with near real-time support by telemedicine | Classification of type of heart failure by will be tested on day 0 (time of study inclusion)
  Comparison of classification of type of heart failure (reduced ejection fraction, mildly reduced ejection fraction or preserved ejection fraction) by the telemedicine approach compared to reference imaging.
  reference echocardiography by cardiologist
Evaluation of volume status with echocardiography by nurses with near real-time support by telemedicine | Evaluation of volume status will be tested on day 0 (time of study inclusion)
  Comparison of volume status (classified individually by a score based on dimension and respiratory variation of the inferior vena cava, visual and Doppler echocardiography and quantification of pleural effusion) by the telemedicine approach compared to reference imaging by cardiologist

CONTACTS AND LOCATIONS:
Overall Officials: Havard Dalen, MD, PhD, Principal Investigator — Helse Nord-Trøndelag HF
Locations (1):
- Levanger Hospital, Levanger, Norway